CLINICAL TRIAL: NCT00004399
Title: Randomized Study of Nimodipine Versus Magnesium Sulfate in the Prevention of Eclamptic Seizures in Patients With Severe Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 199/13249; UU-FDR001061; BCM-FDR001061
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-01

CONDITIONS: Pre-eclampsia
Keywords: cardiovascular and respiratory diseases; hypertensive disorder; pre-eclampsia; rare disease
MeSH Terms: conditions — Pre-Eclampsia; Respiratory Tract Diseases; Hypertension; Rare Diseases | interventions — Magnesium Sulfate; Nimodipine

INTERVENTIONS:
Drug: magnesium sulfate
Drug: nimodipine

SUMMARY:
OBJECTIVES:

I. Determine the effectiveness of nimodipine versus magnesium sulfate in the prevention of eclamptic seizures in patients with severe preeclampsia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, international, multicenter study. Patients are randomized to receive either nimodipine or magnesium sulfate.

Arm I: Patients receive nimodipine by mouth every 4 hours. Treatment is continued until 24 hours post-partum.

Arm II: Patients receive a loading dose of magnesium sulfate IV for 20 minutes, followed by continuous infusion of magnesium sulfate. Treatment is continued until 24 hours post-partum.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Histologically diagnosed severe preeclampsia at risk for eclamptic convulsions with the following criteria:
* Blood pressure greater than 160/110 mmHg OR Mean arterial pressure of 126 mmHg
* Proteinuria greater than 5 g/24 hr
* Epigastric pain OR Right upper quadrant pain AST/ALT greater than 70 U/L
* Severe headache and/or scotomata
* Thrombocytopenia as evidenced by: Platelet count less than 100,000/mm3 Disseminated intravascular coagulation Microangiopathic hemolytic anemia Oliguria (less than 400 mL/day or 30 mL/hr)
* Pulmonary edema

--Prior/Concurrent Therapy--

* No prior/concurrent magnesium sulfate or dihydropyridine agents
* No other concurrent antiseizure medications

--Patient Characteristics--

* Age: Not specified
* Performance status: Not specified
* Hematopoietic: See Disease Characteristics
* Hepatic: See Disease Characteristics
* Renal: No severe renal failure See Disease Characteristics
* Cardiovascular: No history of angina or myocardial infarction No cardiac dysfunction No history or sign of congestive cardiac failure No arrhythmia with ventricular rate less than 60 bpm See Disease Characteristics
* Pulmonary: See Disease Characteristics

--Other:--

* No severe mental or physical disorder that may affect therapy
* Not allergic to drugs with chemical structure similar to nimodipine or magnesium sulfate
* No evidence of fetal distress or fetal anomalies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 1995-09; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Michael Anthony Belfort, Study Chair — University of Utah